CLINICAL TRIAL: NCT03585608
Title: Effect of Neck Extension on Optic Nerve Sheath Diameter in Patients Undergoing Palatoplasty
Brief Title: Optic Nerve Sheath Diameter in Patients Undergoing Palatoplasty
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, Professor, Asan Medical Center
Other Study IDs: 2018-0756
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Neck extension — The neck extension is routine posture during palatoplasty. We will evaluate the change in optic nerve sheath diameters before and after neck extension.

SUMMARY:
The purpose of this study is to evaluate the change of the optic nerve sheath diameter according to the change of the neck position in pediatric patients undergoing palatoplasty.

DETAILED DESCRIPTION:
Palatoplaty is performed under neck extension in patients with cleft palate. The purpose of this study is to evaluate the effect of neck extension on the ultrasonographic optic nerve sheath diameter during palatoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone a palatoplasty with cleft palate and who are 6 months or older and under 24 months
* Patients who agree to voluntarily participate in this study
* Patients with ASA class 1-2

Exclusion Criteria:

* History of diagnosis of neurologic or ophthalmic disease
* History of neurosurgery or ophthalmic surgery
* Patients who refused to participate in clinical studies

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who have undergone a palatoplasty with cleft palate and who are 6 months or older and under 24 months
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Difference in optic nerve sheath diameter | 10 minutes after neck extension
  Difference between the optic nerve sheath diameter measured during supine position without neck extension and the optic nerve sheath diameter measured during supine position with neck extension in patients undergoing palatoplasty

SECONDARY OUTCOMES:
Difference in optic nerve sheath diameter | at end of surgery with the neck extended
  Difference between the optic nerve sheath diameter measured during supine position without neck extension and the optic nerve sheath diameter measured during supine position with neck extension in patients undergoing palatoplasty

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD,PhD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan medical Center, Seoul
  - Young-Kug Kim, Seoul